CLINICAL TRIAL: NCT04479280
Title: Evaluation of the Role of Sonoclot Signature in Assessment of Coagulopathy in Critically Ill COVID 19 Patients
Brief Title: Evaluation of Coagulopathy in Critically Ill COVID-19 Patients.
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Azza Abdelaal, lecturer of clinical pathology, Assiut University
Other Study IDs: 17300446
Record Dates: First submitted 2020-07-19; First posted 2020-07-21 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Coagulation Disorder
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Covid19 positive patients
  Interventions: Device: Sonclot Coagulation and platelet function Analyzer SCP1, Sienco, USA
- Covid19 negative patients
  Interventions: Device: Sonclot Coagulation and platelet function Analyzer SCP1, Sienco, USA

INTERVENTIONS:
Device: Sonclot Coagulation and platelet function Analyzer SCP1, Sienco, USA — studying coagulation disorders in COVID19 critically ill patients

SUMMARY:
Novel coronavirus disease 19 (COVID-19) is caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), this pneumonia was first emerged in December 2019 in Wuhan, China and rapidly spread around the world .

Coagulopathy is one of the most significant prognostic factors in patients with COVID-19 and is associated with increased mortality and admission to critical care. Most observed coagulopathy in patients hospitalized with COVID-19 (COVID-19-associated coagulopathy) is characterized by increased D-dimer and fibrinogen levels. 71% of patients who did not survive hospitalization reported to have developed disseminated intravascular coagulation

ELIGIBILITY:
Inclusion Criteria:

* COVID 19 critically ill patients

Exclusion Criteria:

* any critical illness not related to COVID 19

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who are suspected to be COVID 19 infection
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-08-16 (Actual); Study Completion 2020-08-16 (Actual)

PRIMARY OUTCOMES:
clot rate formation | 30 minutes
  measuring how rapid the sample will get clotted

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt